CLINICAL TRIAL: NCT06721936
Title: Genitourinary Syndrome of Menopause Induced by Breast Cancer Treatments: A Randomized Clinical Trial Protocol Comparing Multimodal Pelvic Floor Physiotherapy and Frac-tional CO2 Laser Therapy (PILME Study).
Brief Title: Genitourinary Syndrome of Menopause in Breast Cancer
Acronym: PILME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Full Professor, University of Alcala
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/1/012
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Genitourinary Syndrome of Menopause (GSM); Breast Cancer Female
Keywords: Breas cancer; Cost-effectiveness; Dyspareunia; Genitourinary syndrome of menopause; Laser therapy; Menopause; Physiotherapy; Quality of life
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser CO2 Therapy group (Active Comparator): Participants in this group will undergo three treatment sessions using the Monalisa Touch CO2 fractional laser, administered by a senior gynaecologist (MD3) on an outpatient basis, once a month for three consecutive months. Each session will last approximately 15 minutes and will be performed without anaesthesia
  Interventions: Device: Laser CO2 Therapy group
- Multimodal pelviperineal physioterapy group (Experimental): Participants in this group will attend eight personalized sessions of multimodal PPT, each lasting 50-60 minutes, administered once a week the six first sessions, and the last 2 sessions, one session every two weeks. The multimodal PPT protocol includes: 1) Pelvic Floor Muscle Training (PFMT); 2) Non-Ablative Radiofrequency Therapy (Model: RNG, INDIBA); 3) Therapeutic Pelvic Health Education.
  Interventions: Combination Product: Multimodal pelviperineal physioterapy group

INTERVENTIONS:
Combination Product: Multimodal pelviperineal physioterapy group — The multimodal PPT protocol includes:
  Pelvic Floor Muscle Training (PFMT): This component includes techniques to raise awareness of the pelvic floor, incorporating both manual and instrumental intravaginal techniques.
  Non-Ablative Radiofrequency Therapy (Model: RNG, INDIBA): Applied during all eight sessions, with each session lasting 25 minutes.
  Therapeutic Pelvic Health Education: Designed to empower participants with knowledge about their condition and the pelvic-perineal area. This educational intervention aims to enhance understanding, promote self-care, and encourage behaviours that alleviate symptoms associated with GSM
  Arms: Multimodal pelviperineal physioterapy group
Device: Laser CO2 Therapy group — The fractional laser application will be delivery with the following probes:
  90° Probe for Incontinence: Maximum power of 40W; 360° Probe for Vaginal Atrophy: Maximum power of 40W and Right-Angle Probe for Vulvar Atrophy: Maximum power of 24W.
  Arms: Laser CO2 Therapy group

SUMMARY:
This randomized, single-blind clinical trial will compare the effectiveness of multimodal pelvic floor physiotherapy (PPT) and fractional CO2 vaginal laser therapy in reducing genitourinary syndrome of menopause (GSM) symptoms among breast cancer (BC) survivors. GSM, induced by cancer treatments, is common in BC survivors due to hormonal deprivation, and effective non-hormonal treatments are needed. The study will enroll 210 women diagnosed with GSM following BC treatment, who will be randomly assigned to either three sessions of CO2 vaginal laser therapy or eight sessions of multimodal PPT, which includes pelvic floor muscle training, vaginal non-ablative radiofrequency, education, and moisturizers. Primary outcomes will include perineal pain, sexual function, and health-related quality of life (HRQoL), with assessments at baseline, post-intervention, and at 3, 6, and 12 months. The hypothesis is that multimodal PPT will lead to greater improvements in pelvic pain, muscle function, and sexual health, with sustained benefits over time. This trial aims to provide evidence for non-invasive, non-hormonal treatments to manage GSM in BC survivors, filling a significant therapeutic gap.

DETAILED DESCRIPTION:
Background: Genitourinary syndrome of menopause (GSM) induced by breast cancer (BC) treatments is highly prevalent among BC survivors due to the abrupt hor-monal deprivation caused by oncological therapies. Given the contraindication of hor-monal treatments in this population, there is a critical need for effective non-hormonal alternatives to alleviate GSM symptoms.

Objectives: This study aims to compare the effectiveness of multimodal pelvic floor physiotherapy (PPT)-comprising pelvic floor muscle training, vaginal non-ablative radiofrequency, pelvic health education, and vaginal moisturizers-against fractional CO2 vaginal laser therapy in reducing GSM symptoms among BC survivors.

Methods: A randomized, single-blind clinical trial will be conducted with 210 women diagnosed with GSM after undergoing BC treatment. Participants will be ran-domly assigned (1:1) to receive either three sessions of CO2 vaginal laser therapy or eight face-to-face sessions of multimodal PPT. Assessments will be performed at base-line, immediately after the intervention, and at 3-, 6-, and 12- months post-intervention. Primary outcomes will include perineal pain, sexual function, and health-related quality of life (HRQoL). Additionally, a cost-effectiveness analysis will be conducted to evaluate the costs of each intervention relative to the changes in clinical outcomes, and any ad-verse effects will be monitored throughout the study.

Results: It is hypothesized that women undergoing multimodal PPT will show greater reductions in pelvic pain and improvements in pelvic floor muscle strength, endurance, and relaxation compared to those receiving CO2 laser therapy, alongside enhanced sexual function and HRQoL. These improvements are expected to be sus-tained in the short and medium term through continued adherence to home exercises and educational strategies.

Conclusions: This study aims to provide evidence for novel, non-invasive, and non-hormonal treatment strategies to manage GSM in BC survivors, addressing an important gap in the therapeutic landscape for this population.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors diagnosed with GSM as a result of cancer treatment
* Vaginal Health Index (VHI) score of ≤ 15.

Exclusion Criteria:

* History of conservative treatment or surgery for pelvic floor dysfunction or GSM
* Currently undergoing chemotherapy, or have undergone BC surgery but have not received chemotherapy or hormonal treatment.
* Presence of concomitant or systemic diseases that could interfere with the proposed treatments, such as a recurrence of the oncological process, active or recurrent untreated urinary tract infections, hematuria, or cognitive impairments that hinder the participant's ability to comprehend study information, respond to questionnaires, provide informed consent, or fully participate in the study.

Min Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function (FSFI) | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  The FSFI is a 19-item questionnaire that evaluates sexual function across six domains: de-sire, arousal, lubrication, orgasm, satisfaction, and pain. Each domain is scored from 0 to 5, with higher scores indicating better sexual function. The total FSFI score ranges from 2 to 36, with higher scores reflecting improved sexual function.
Subjective Pelvic Perineal Pain Intensity | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Measured using a 100-mm horizontal Visual Analog Scale (VAS), with "no pain" on the left and "worst imaginable pain" on the right.
Health-Related Quality of Life (HRQoL) | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  This 40-item questionnaire evaluates HRQoL across four general domains (physical, emo-tional, social, and functional well-being), along with two specific subscales: breast cancer (9 items) and arm symptoms (4 items). The scores for the BC subscale (BCS) and arm subscale range from 0 to 56. The Trial Outcome Index (TOI), a key measure, is the sum of the BCS and the physical and functional well-being subscales, with scores ranging from 0 to 92. The total FACT-B score ranges from 0 to 144, where higher scores indicate better HRQoL.

SECONDARY OUTCOMES:
Vaginal Health Index (VHI) | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  This index evaluates five key aspects of vaginal health: elasticity, epithelial integrity, pH, hydration, and fluid volume. Each component is scored from 1 to 5, with lower scores in-dicating poorer vaginal health. A VHI score of ≤15 indicates vaginal atrophy.
Impact of Vaginal Symptoms | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  The Day-to-Day Impact of Vaginal Aging (DIVA) questionnaire assesses the impact of vulvovaginal symptoms in postmenopausal women across four domains: activities of daily living, emotional well-being, sexual functioning, and self-concept/body image. The ques-tionnaire consists of 22 items, each scored on a scale from 0 to 4. The score for each domain is calculated by averaging the scores of its items, with higher scores indicating a greater impact of vaginal symptoms.
Pelvic Floor Dysfunction Symptoms | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Assessed using the Spanish version of the Pelvic Floor Distress Inventory-Short Form (PFDI-20), which consists of 20 questions across three subscales: prolapse, anal, and uri-nary symptoms. The total score ranges from 0 to 300, with higher scores indicating greater distress.
Treatment Satisfaction | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Satisfaction with the treatment will be assessed using a numerical verbal scale ranging from 0 to 10, where 0 represents no satisfaction and 10 indicates excellent satisfaction. This evaluation will begin with assessment A1.
Pelvic Floor Muscle Tone | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Measured using vaginal dynamometry with the Pelvimetre™ (Phenix Vivaltis, Montpel-lier, France). For the assessment, the participant will be in lithotomy position, and the tone of the pelvic floor muscles will be considered when the vaginal device is inserted, and the participant perceives that her muscles are relaxed.
Pelvic Floor Muscle Strength | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Measured using vaginal dynamometry with the Pelvimetre™ (Phenix Vivaltis, Montpel-lier, France). The participant, in the lithotomy position, will perform three maximum contractions of the pelvic floor muscles. The average value of the three contractions will be considered.
Pelvic Floor Muscle Contraction | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  Three maximum pelvic floor muscle contractions will be requested in lithotomy position, and the distance of the urogenital hiatus will be assessed using transperineal ultrasound (Mindray M7, Shenzhen, China).
Pelvic Floor Elasticity | Baseline (before intervention) (A0); immediately after completing the intervention (A1), and at 3 months (A2), 6 months (A3), and 12 months (A4) following A1.
  In the lithotomy position, an inspiratory apnea Valsalva maneuver will be requested, and the distance of the urogenital hiatus will be assessed using transperineal ultrasound (Mindray M7, Shenzhen, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Torres-Lacomba M, Hernandez-Iglesias CM, Del Valle-Rubido C, Navarro-Brazalez B, Rangel-de la Mata P, Lorenzo-Gallego L, Sanchez-Sanchez B, Salvador-Osuna M, Lazaro-Carrasco de la Fuente J. Genitourinary syndrome of menopause induced by breast cancer treatments: a randomised clinical trial protocol comparing multimodal pelvic floor physiotherapy and fractional CO2 laser therapy (PILME study). BMJ Open. 2025 Nov 27;15(11):e104711. doi: 10.1136/bmjopen-2025-104711. PMID 41309480